CLINICAL TRIAL: NCT05354401
Title: Use of Heated Humidified High Flow Nasal Cannula Oxygen in Obstructive Sleep Apnea in Adolescents With Obesity and Complex Medical Conditions
Brief Title: Heated Humidified High Flow Nasal Cannula Oxygen in Obstructive Sleep Apnea in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1000054076
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Obstructive Sleep Apnea (Moderate to Severe); Central Sleep Apnea
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese (Active Comparator): Obese subjects ages 10-18 years with OSA will be recruited from sleep clinic. As per standard clinic care, once a subject is diagnosed with OSA on a PSG they are reviewed in sleep clinic to discuss CPAP therapy. Families will be approached to participate in this study during the subject's regularly scheduled clinical visit. Obese subjects meeting eligibility criteria will be recruited from the sleep clinic. The patients agreeing to CPAP therapy will be invited to take part in the study.
  Interventions: Other: HHF
- CMC (Active Comparator): As per current standard clinical care, CMC diagnosed with moderate to severe OSA following a clinically indicated baseline PSG who have had a previous adenotonsillectomy or who are not considered candidates for surgery are reviewed in sleep clinic to discuss the prescription of CPAP for OSA. CMC subjects' meeting eligibility criteria will be recruited from the sleep clinic. The patients agreeing to CPAP therapy will be invited to take part in this study.
  Interventions: Other: HHF

INTERVENTIONS:
Other: HHF — HHF is an integrated flow generator that delivers heated and humidified air or oxygen at high flow rates via a soft nasal cannula using an open circuit. HHF via the Fisher and Paykel myAIRVO 2 device will be initiated as per The Hospital for Sick Children's sleep laboratory standard protocol by a sleep technician or respiratory therapist (RT) during an overnight polysomnography. Nasal prongs will be selected that are less than fifty percent of the subject's nares. The lowest flow rate of HHF will be selected and titrated upwards until clinical effect is achieved, to a maximum flow of 60L/minute, as per standard clinical care.

SUMMARY:
The research study is being done to test heated humidified high-flow air (HHF), as a treatment for OSA.

ELIGIBILITY:
OBESE SUBJECTS:

Inclusion Criteria:

* Obesity, defined as a BMI > 95th percentile for age and gender
* Age 10 through 18 years
* Informed consent with assent in accordance with the institutional policies (institutional IRB approval) must be signed by the patient's legally authorized guardian acknowledging written consent to join the study
* Moderate-severe OSA or Central Sleep Apnea (CSA) as defined by OAHI or CAHI

Exclusion Criteria:

* Patients with other neurological problems, including but not limited to neurocutaneous disorders such as neurofibromatosis or tuberous sclerosis
* Obesity due to other diseases and syndromes (e.g. Prader-Willi syndrome)
* Pregnancy
* Currently unwell, hospitalized or recent viral/bacterial infection in the previous 4 weeks
* Adenoidal and/or tonsillar hypertrophy which may be amenable to surgical intervention to help alleviate OSA
* Patients with severe respiratory distress
* Patients with increased risk of pneumothorax including but not limited to previous pneumothorax, bronchiectasis or severe untreated asthma.

CHILDREN WITH MEDICAL COMPLEXITY SUBJECTS:

Inclusion Criteria:

* CMC recently diagnosed with moderate to severe OSA or CSA requiring CPAP therapy
* 0-18 years of age
* Informed consent with assent in accordance with the institutional policies (institutional IRB approval) must be signed by the patient's legally authorized guardian acknowledging written consent to join the study

Exclusion Criteria:

* Current upper respiratory tract infection
* Subjects who are receiving oxygen therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI) with HHF compared to the change in AHI with CPAP | week 1-4
  Determine whether a participant's AHI changes with HHF vs CPAP

SECONDARY OUTCOMES:
Comparative COMFORT scales with HHF and CPAP. | week 1-4
  Determine whether COMFORT scale scores differ between HHF and CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, BMEDSci, MBBCH, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Fishman H, Al-Shamli N, Sunkonkit K, Maguire B, Selvadurai S, Baker A, Amin R, Propst EJ, Wolter NE, Eckert DJ, Cohen E, Narang I. Heated humidified high flow nasal cannula therapy in children with obstructive sleep apnea: A randomized cross-over trial. Sleep Med. 2023 Jul;107:81-88. doi: 10.1016/j.sleep.2023.04.017. Epub 2023 Apr 21. PMID 37148831